CLINICAL TRIAL: NCT07281079
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Orally Administered NNZ-2591 Compared With Placebo in Pediatric Participants With Phelan-McDermid Syndrome
Brief Title: A Study of NNZ-2591 in Pediatric Participants With Phelan-McDermid Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEU-2591-PMS-301
Record Dates: First submitted 2025-11-13; First posted 2025-12-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Phelan-McDermid Syndrome
Keywords: Phelan McDermid Syndrome; NEU-2591-PMS-301; NNZ-2591; Neuren
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome | interventions — cyclo-L-glycyl-L-2-allylproline

STUDY DESIGN:
Intervention Model Description: Phase 3, randomized, double-blind, parallel-group (2-arm), placebo-controlled, multicenter study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) This is a double-blind study in which pediatric participants, caregivers, investigators, and the sponsor are blinded to study drug for the duration of study. Dose escalation, dose modification, and treatment discontinuation will be performed in a blinded manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNZ-2591 Arm (Experimental): The total duration of this study for each participant will be up to approximately 17 to 19 weeks.
  Participants will be randomized in a 1:1 ratio to receive orally administered NNZ-2591 during the 13-week Treatment Period.
  Interventions: Drug: NNZ-2591
- Placebo Arm (Placebo Comparator): The total duration of this study for each participant will be up to approximately 17 to 19 weeks.
  Participants will be randomized in a 1:1 ratio to receive orally administered placebo matching NNZ-2591 during the 13-week Treatment Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNZ-2591 — The study drug will be administered twice daily orally.
  Arms: NNZ-2591 Arm
Drug: Placebo — The study drug will be administered twice daily orally.
  Arms: Placebo Arm

SUMMARY:
This Phase 3, randomized, double-blind, parallel-group (2-arm), placebo-controlled, multicenter study will evaluate the efficacy and safety of NNZ-2591 compared to placebo in pediatric participants with Phelan- McDermid Syndrome.

DETAILED DESCRIPTION:
After providing informed consent/assent, pediatric participants with Phelan-McDermid syndrome ages 3-12 years of age will enter the 4-week Screening Period and undergo assessments for eligibility, baseline characteristics and symptom severity.

Once eligibility is confirmed, participants will be randomized in a 1:1 ratio to receive either orally administered NNZ-2591 or matching placebo during the 13-week Treatment Period. Subsequently, a 2-week safety follow-up period will occur immediately after the completion of the Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female pediatric participants with Phelan-McDermid syndrome ages 3 to 12 years (inclusive) at the time of signing the informed consent.
2. Clinical diagnosis of Phelan-McDermid syndrome with a documented disease-causing genetic abnormality of SHANK3.
3. Body weight ≥ 10 kg at Screening.
4. Participants with a PMSA-S overall score ≥ 3 at the Screening and Baseline visits.
5. Not actively undergoing regression or loss of skills.

Exclusion Criteria:

1. Use of exclusionary medication or unstable treatment regimens of acceptable concomitant medications as required by the protocol.
2. Current treatment with more than 3 allowable psychotropic medications.
3. Participants with seizures must be controlled on no more than 2 anticonvulsant medications (not counting rescue medications).
4. Psychotropic medications or any other medication used for a chronic illness (not including antibiotics, pain relievers, anti-diarrheals, and laxatives) with doses and dosing regimen that have not been stable for at least 4 weeks before Screening. If the treatment was discontinued, the discontinuation must have occurred no fewer than 2 weeks before the start of Screening.
5. Any intercurrent seizures in the past 6 months and /or more than 1 seizure in the past 12 months. •A single febrile seizure in the 6 months prior to screening is allowable if no rescue medication was required.
6. Abnormal liver function laboratory results during the Screening period, as defined by the protocol
7. Abnormal QT interval on Screening ECG as defined by the protocol.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy of NNZ-2591 compared with placebo as measured by the Phelan-McDermid Syndrome Assessment of Change (PMSA-C) overall score. | Week 13
  Efficacy of NNZ-2591 compared with placebo as measured by the Phelan-McDermid Syndrome Assessment of Change (PMSA-C) overall score. The PMSA-C scores range from 1 to 7 with 1 indicating very much improved and 7 indicating very much worse.
Efficacy of NNZ-2591 compared with placebo as measured by the change from baseline in the Vineland Adaptive Behavior Scales-3, Interview version (Vineland-3) receptive communication subdomain raw score. | Week 13
  Efficacy of NNZ-2591 compared with placebo as measured by the change from baseline in the Vineland Adaptive Behavior Scales-3, Interview version (Vineland-3) receptive communication subdomain raw score. A higher raw score for the receptive communication subdomain indicates better adaptive behavior.

SECONDARY OUTCOMES:
Efficacy of NNZ-2591 compared with placebo as measured by the Caregiver Impression of Change (CIC) overall score. | Week 13
  Efficacy of NNZ-2591 compared with placebo as measured by the Caregiver Impression of Change (CIC) overall score. The CIC scores range from 1 to 7 with 1 indicating very much improved and 7 indicating very much worse.
Efficacy of NNZ-2591 compared with placebo as measured by the Phelan-McDermid Syndrome Assessment of Change (PMSA-C) domain scores. | Week 13
  Efficacy of NNZ-2591 compared with placebo as measured by the Phelan-McDermid Syndrome Assessment of Change (PMSA-C) domain scores. The PMSA-C domain scores range from 1 to 7 with 1 indicating very much improved and 7 indicating very much worse.
Efficacy of NNZ-2591 compared with placebo as measured by the Caregiver Impression of Change (CIC) domain scores. | Week 13
  Efficacy of NNZ-2591 compared with placebo as measured by the Caregiver Impression of Change (CIC) domain scores. The CIC scores range from 1 to 7 with 1 indicating very much improved and 7 indicating very much worse.
Efficacy of NNZ-2591 compared with placebo as measured by the change from baseline in Phelan-McDermid Syndrome Assessment of Severity (PMSA-S) domain scores. | Week 13
  Efficacy of NNZ-2591 compared with placebo as measured by the change from baseline in Phelan-McDermid Syndrome Assessment of Severity (PMSA-S) domain scores. The PMSA-S scores range from 1 to 7 with 1 indicating typical for age, not at all impaired and 7 among the most severely impaired.
Efficacy of NNZ-2591 compared with placebo as measured by the change from baseline in PMSA-S overall score. | Week 13
  Efficacy of NNZ-2591 compared with placebo as measured by the change from baseline in PMSA-S overall score. The PMSA-S scores range from 1 to 7 with 1 indicating typical for age, not at all impaired and 7 among the most severely impaired.
Efficacy of NNZ-2591 compared with placebo as measured by the change from baseline in PMS Clinician Domain Specific Rating Scale (PMS-DSRS) scores. | Week 13
  Efficacy of NNZ-2591 compared with placebo as measured by the change from baseline in PMS Clinician Domain Specific Rating Scale (PMS-DSRS) scores. The PMS-DSRS scores range from 0 to 4 with 0 indicating Symptom Not Present and 4 indicating Very Severe.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Neuren PMS-301 Site#111, San Rafael, California
  - Neuren PMS-301 Site#109, Chevy Chase, Maryland

IPD SHARING:
Plan to Share IPD: No